CLINICAL TRIAL: NCT02804698
Title: Tools And Practices To Decrease CVD And Complications In The Diabetic Population Of Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: El Colegio de Sonora (Unknown)
Responsible Party: Principal Investigator, Cecilia B Rosales, Professor, Public Health / Assistant Dean, Phoenix Campus, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1508040144
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Diabetes; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meta Salud Diabetes-Intervention (Experimental): 1. Attend the thirteen weekly educational classes and physical activity group (prior physician approval) that are part of the Meta Salud Diabetes program.
  2. Allow the research staff to collect your cholesterol, glucose, A1c, triglyceride levels, as well as your blood pressure, height, weight, and waist and hip circumference.
  3. Respond to a survey about your nutrition and physical activity habits on three separate occasions (at the start of the 13-week program, just after you finish the program, and nine months after you finish the program).
  4. You may also be invited to participate in a follow-up interview, where you will be asked about your experience during and after the Meta Salud Diabetes program.
  Interventions: Behavioral: Education intervention
- Meta Salud Diabetes-Comparison Group (No Intervention): 1. Allow the research staff to collect your cholesterol, glucose, A1c, triglyceride levels, as well as your blood pressure, height, weight, and waist and hip circumference.
  2. Respond to a survey about your nutrition and physical activity habits on three separate occasions (you will answer the first survey as soon as you finish reading and agree to participate by signing this form, the second survey will be three months from now, and the third survey will be 12 months from now).

INTERVENTIONS:
Behavioral: Education intervention — 13-week educational and physical activity intervention
  Arms: Meta Salud Diabetes-Intervention

SUMMARY:
This project will look to improve standards of care for diabetic patients by evaluating a program that supports participants in making healthy lifestyle changes.

The program consists of 13 educational sessions that contain information about the prevention and care of diabetes and cardiovascular disease, physical activity, nutrition, community health and emotional well being.

DETAILED DESCRIPTION:
Researchers propose to address extremely high rates of cardiovascular disease morbidity and mortality in Sonora, Mexico through use of an evidence-based community health worker intervention for adult patients with diabetes who receive care at health centers operated by the Secretaría de Salud, an office of the Mexican government. Researchers will conduct a cluster-randomized trial with a total of 400 patients at 20 health centers to understand whether the 13-week educational intervention, Meta Salud Diabetes, can effectively reduce clinical, behavioral, and psychosocial risk for cardiovascular disease among adults with diabetes. Researchers will also conduct an implementation study that will consist of systematic engagement of local, state and national decision makers to identify barriers, facilitators, and strategies to adopt and integrate community health worker-led cardiovascular disease prevention interventions throughout the 209 health centers in Sonora.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥18 years old
* have been diagnosed with controlled or uncontrolled diabetes

Exclusion Criteria:

* < than 18 years of age
* not diagnosed with diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Framingham cardiovascular disease risk | 12 months
  Risk Scores estimate the probability that a person will develop CVD

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia B Rosales, MD, MS, Principal Investigator — University of Arizona
Locations (1):
- Ministry of Health, Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aceves B, Denman CA, Ingram M, Torres JF, Nuno T, Garcia DO, Madhivanan P, Rosales CB. Testing Scalability of a Diabetes Self-Management Intervention in Northern Mexico: An Ecological Approach. Front Public Health. 2021 Aug 18;9:617468. doi: 10.3389/fpubh.2021.617468. eCollection 2021. PMID 34490173
- [Derived] Aceves B, Ruiz M, Ingram M, Denman C, Garcia DO, Madhivanan P, Rosales C. Mental health and diabetes self-management: assessing stakeholder perspectives from health centers in Northern Mexico. BMC Health Serv Res. 2021 Feb 25;21(1):177. doi: 10.1186/s12913-021-06168-y. PMID 33632205
- [Derived] Bell ML, Rabe BA. The mixed model for repeated measures for cluster randomized trials: a simulation study investigating bias and type I error with missing continuous data. Trials. 2020 Feb 7;21(1):148. doi: 10.1186/s13063-020-4114-9. PMID 32033617
- [Derived] Ingram M, Denman CA, Cornejo-Vucovich E, Castro-Vasquez MDC, Aceves B, Ocejo AG, de Zapien JG, Rosales C. The Meta Salud Diabetes Implementation Study: Qualitative Methods to Assess Integration of a Health Promotion Intervention Into Primary Care to Reduce CVD Risk Among an Underserved Population With Diabetes in Sonora, Mexico. Front Public Health. 2019 Nov 15;7:347. doi: 10.3389/fpubh.2019.00347. eCollection 2019. PMID 31803710
- [Derived] Sabo S, Denman Champion C, Bell ML, Cornejo Vucovich E, Ingram M, Valenica C, Castro Vasquez MDC, Gonzalez-Fagoaga E, Geurnsey de Zapien J, Rosales CB. Meta Salud Diabetes study protocol: a cluster-randomised trial to reduce cardiovascular risk among a diabetic population of Mexico. BMJ Open. 2018 Mar 12;8(3):e020762. doi: 10.1136/bmjopen-2017-020762. PMID 29530914